CLINICAL TRIAL: NCT07229807
Title: A Phase 3 Study of ZSP1273 in Otherwise Healthy Children 2-11 Years Old With Influenza A
Brief Title: Efficacy and Safety of ZSP1273 in Children 2-11 Years Old With Influenza A
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZSP1273-25-20
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Influenza a
MeSH Terms: interventions — ZSP1273; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZSP1273 (Experimental)
  Interventions: Drug: ZSP1273
- Oseltamivir (Active Comparator)
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: ZSP1273 — Oral
  Arms: ZSP1273
Drug: Oseltamivir — Oral
  Arms: Oseltamivir

SUMMARY:
This trial is conducted in China. The aim of the trial is to investigate safety and efficacy of ZSP1273 granules

ELIGIBILITY:
Inclusion Criteria:

1. Participants and their guardians who are able to understand the study and comply with all study procedures, and willing to provide written informed consent/assent prior to the predose examinations appropriately.
2. Male or female participants aged ≥ 2 to ≤11 years at the time of signing the informed consent form.
3. Participants with a diagnosis of influenza virus infection confirmed by all of the following:

   1. Positive rapid antigen test (RAT) for influenza with nasal or throat swabs;
   2. The time interval between the onset of symptoms and enrollment is 48 hours or less;
   3. Fever ≥ 38ºC (axillary temperature); and at least one following respiratory symptoms associated with influenza virus infection is present

Exclusion Criteria:

1. Participants with severe influenza virus infection；
2. Participants with any medical history in gastrointestinal that interferes with the absorption of drugs；
3. Immunodeficiency,including malignant tumor,organ or marrow transplant,human immunodeficiency virus [HIV] infection,or patients receiving immunosuppressant therapy 3 months prior to enrollment；
4. Have received any other investigational products within 3 months prior to dosing；
5. Positive urine pregnancy test；
6. Participants with concurrent infections requiring antimicrobial therapy；
7. Participants who are considered inappropriate for the study by the investigator.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Alleviation of Symptoms | DAY1~DAY15
  Participants assessed the severity of influenza-associated symptoms

SECONDARY OUTCOMES:
Plasma concentrations of ZSP1273 | DAY1~5
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | DAY1~15

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No